CLINICAL TRIAL: NCT04373343
Title: Pilot Investigation of a Novel Therapeutic Intervention for Food Addiction: Food Addiction Clinical Treatment (FACT) Program
Brief Title: Food Addiction Clinical Treatment Program
Acronym: FACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB00053663
Record Dates: First submitted 2020-04-21; First posted 2020-05-04 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-01

CONDITIONS: Food Addiction
Keywords: Obesity Associated Disorder; Binge Eating; Weight, Body
MeSH Terms: conditions — Food Addiction; Bulimia; Body Weight

STUDY DESIGN:
Intervention Model Description: Males and females meeting criteria for severe food addiction and interested in completing 16 week pilot treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 16-week Food Addiction Clinical Treatment (FACT) Program (Other): 16-week Food Addiction Clinical Treatment (FACT) Program, first session will be 120 mins, all subsequent sessions will be 90 mins. Treatment will be led, at a minimum, by a full licensed psychologist
  Interventions: Behavioral: 16-week Food Addiction Clinical Treatment (FACT) Program

INTERVENTIONS:
Behavioral: 16-week Food Addiction Clinical Treatment (FACT) Program — 16-week Food Addiction Clinical Treatment (FACT) Program, first session will be 120 mins, all subsequent sessions will be 90 mins. Treatment will be led, at a minimum, by a full licensed psychologist

SUMMARY:
The purpose of this current study is to establish the feasibility of, and preliminary support for, a clinical treatment program utilizing interventions from various empirically supported treatments for obesity-related eating disorders and substance use disorders

DETAILED DESCRIPTION:
To establish the feasibility of recruiting, enrolling, and treating individuals who meet criteria for FA in a group behavioral intervention for 16 weeks. Data from the current study will be used for the purposes of further exploration of the FACT program in a larger randomized controlled trial. We hypothesize the study will demonstrate the feasibility of evaluating this treatment in future studies

ELIGIBILITY:
Inclusion Criteria:

* Age > 25
* BMI >25
* YFAS > 6/11 (severe range)
* willing to commit to a 16 week group therapy program from 4 - 5:30 pm on Thursdays in Winston-Salem, NC
* English speaking

Exclusion Criteria:

* Current participation in professional weight loss program and unwillingness to suspend it for 16 weeks during treatment
* obesity medications with exception of diabetes medication with weight loss benefit (ie metformin),
* current nicotine use or substance use disorder (based on meeting the clinical cutoff for the Alcohol Use Disorders Identification Test and/or Cannabis Use Disorder Identification Test
* history of weight loss surgery,
* current/history of severe mental illness (> 3 psychiatric hospitalizations since age 18,
* schizoaffective disorder, bipolar disorder, psychotic disorder, or personality disorder),
* current/history of lithium, abilify, saphris, vraylor, clozaril, latuda, zyprexa, seroquel, risperdal, or Geodon,
* current pregnancy or breastfeeding,
* prior diagnosis of anorexia nervosa, diagnosis of bulimia nervosa in the last 5 years,
* high currents rates of restrictive eating disorder symptoms based on the Eating Disorder Diagnosis Scale (EDDS; (i.e., any endorsement of vomiting or laxative/diuretic use to manage weight and endorsement of fasting or excessive exercise more than 2 or 3 times a week)

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2023-03-21 (Actual); Primary Completion 2023-09-07 (Actual); Study Completion 2023-09-07 (Actual)

PRIMARY OUTCOMES:
Yale Food Addiction Scale 2.0 (YFAS) | pre 16-week intervention
  The YFAS 2.0 is a self-report measure used to assess addictive eating behaviors related to highly processed foods. The YFAS 2.0 consists of 35 items based on the DSM - 5 diagnostic criteria for substance use No Food Addiction = 0-1 symptoms/score Mild Food Addiction = 2 or 3 score Moderate Food Addiction = 4 or 5 score Severe Food Addiction = 6 or higher score
Yale Food Addiction Scale 2.0 (YFAS) | post 16-week intervention
  The YFAS 2.0 is a self-report measure used to assess addictive eating behaviors related to highly processed foods. The YFAS 2.0 consists of 35 items based on the DSM - 5 diagnostic criteria for substance use No Food Addiction = 0-1 symptoms/score Mild Food Addiction = 2 or 3 score Moderate Food Addiction = 4 or 5 score Severe Food Addiction = 6 or higher score
Weight Self-Stigma Questionnaire (WSSQ) | pre 16-week intervention
  WSSQ assesses two aspects of internalized weight stigma: self-devaluation and fear of enacted stigma. It contains 12 items rated on a 5-point Likert scale - Higher scores mean that you experience more shame related to your weight or body shape, while lower scores indicate that you experience less
Weight Self-Stigma Questionnaire (WSSQ) | post 16-week intervention
  WSSQ assesses two aspects of internalized weight stigma: self-devaluation and fear of enacted stigma. It contains 12 items rated on a 5-point Likert scale - Higher scores mean that you experience more shame related to your weight or body shape, while lower scores indicate that you experience less
Patient Health Questionnaire (PHQ-9) with suicide question removed | pre 16-week intervention
  a self-report measure consisting of 9 questions, each aligning with one of the DSM - IV criteria for depression. The Posttraumatic Stress Disorder Checklist (PCL-5) is a 20 item self-report measure that assesses the DSM-5 symptoms of PTSD and is a commonly used tool to screen subjects for PTSD 0-4 Minimal or no depression 5-9 Mild depression 10-14 Moderate 15-19 Moderately severe > 20 Severe
Patient Health Questionnaire (PHQ-9) with suicide question removed | post 16-week intervention
  a self-report measure consisting of 9 questions, each aligning with one of the DSM - IV criteria for depression. The Posttraumatic Stress Disorder Checklist (PCL-5) is a 20 item self-report measure that assesses the DSM-5 symptoms of PTSD and is a commonly used tool to screen subjects for PTSD 0-4 Minimal or no depression 5-9 Mild depression 10-14 Moderate 15-19 Moderately severe > 20 Severe
Generalized Anxiety Disorder (GAD-7) | pre 16-week intervention
  brief self-report assessment of anxiety. The measure consists of 7 items that quickly identify anxiety symptoms and severity - Scores of 5, 10, and 15 are taken as the cut-off points for mild, moderate and severe anxiety, respectively
Generalized Anxiety Disorder (GAD-7) | post16-week intervention
  brief self-report assessment of anxiety. The measure consists of 7 items that quickly identify anxiety symptoms and severity - Scores of 5, 10, and 15 are taken as the cut-off points for mild, moderate and severe anxiety, respectively
Alcohol Use Disorder Identification Test (AUDIT) | pre 16-week intervention
  a self-report measure assessing alcohol consumption, drinking behaviors, and alcohol-related problems. The 10-item scale is used as a screening tool - A score of 8 or more is associated with harmful or hazardous drinking, a score of 13 or more in women, and 15 or more in men, is likely to indicate alcohol dependence
Alcohol Use Disorder Identification Test (AUDIT) | post 16-week intervention
  a self-report measure assessing alcohol consumption, drinking behaviors, and alcohol-related problems. The 10-item scale is used as a screening tool - A score of 8 or more is associated with harmful or hazardous drinking, a score of 13 or more in women, and 15 or more in men, is likely to indicate alcohol dependence
Cannabis Use Disorder Identification Test (CUDIT) | pre 16-week intervention
  a self-report 8 item measure assessing various cannabis use behaviors - Scores can range from 1 to 32, with a cut-off score of 13 indicative of a DSM-IV diagnosis of CUD (dependence)
Cannabis Use Disorder Identification Test (CUDIT) | post 16-week intervention
  a self-report 8 item measure assessing various cannabis use behaviors - Scores can range from 1 to 32, with a cut-off score of 13 indicative of a DSM-IV diagnosis of CUD (dependence)
Sense of Self-Efficacy Scale | pre 16-week intervention
  a questionnaire that measures a participant's level of belief in his or her ability to take the necessary actions to accomplish a goal. It consists of 20 items that assess self-efficacy in the areas of decision-making, coping and social skills, and planning - The scale has a range of scores from 0-90. A higher number on the score represents a higher self-efficacy for exercise.
Sense of Self-Efficacy Scale | post 16-week intervention
  a questionnaire that measures a participant's level of belief in his or her ability to take the necessary actions to accomplish a goal. It consists of 20 items that assess self-efficacy in the areas of decision-making, coping and social skills, and planning - The scale has a range of scores from 0-90. A higher number on the score represents a higher self-efficacy for exercise.
World Health Organization Quality of Life - BREF (WHOQOL-BREF) | pre 16-week intervention
  is a self-report questionnaire assessing the individual's perceptions in the context of their culture and value systems, and their personal goals, standards, and concerns. It consists of 26 items measuring physical health, psychological health, social relationships, and environment - higher scores denote higher quality of life
World Health Organization Quality of Life - BREF (WHOQOL-BREF) | post 16-week intervention
  is a self-report questionnaire assessing the individual's perceptions in the context of their culture and value systems, and their personal goals, standards, and concerns. It consists of 26 items measuring physical health, psychological health, social relationships, and environment - higher scores denote higher quality of life
Physical Fitness Assessment (height) | pre 16-week intervention
  subject's height will be taken using a wall-mounted stadiometer and weight will be taken using a medical-grade scale.
Physical Fitness Assessment (weight) | pre 16-week intervention
  Weight will be measured using the TANITA scale.
Physical Fitness Assessment (weight) | post 16-week intervention
  Weight will be measured using the TANITA scale.
Physical Fitness Assessment (body composition) | pre 16-week intervention
  body composition will be measured using the TANITA scale. This measure provides information about a subject's body fat percentage, body water weight percentage, and lean muscle mass percentage.
Physical Fitness Assessment (body composition) | post 16-week intervention
  body composition will be measured using the TANITA scale. This measure provides information about a subject's body fat percentage, body water weight percentage, and lean muscle mass percentage.
Resting Metabolic Rate | post 16-week intervention
  Resting Metabolic Rate (RMR) will be measured using the CardioCoach or ReeVue (KORR Medical Technologies, Salt Lake City, UT). An RMR measurement uses oxygen consumed at rest to determine a person's caloric requirements for weight loss or maintenance
4-meter timed walk test | pre 16-week intervention
  The 4-meter timed walk test will be used to measure normal gait speed and provide an approximate measure of physical functioning and level of deconditioning. The subject will be instructed to walk at their normal pace through a hallway that has a 4-meter distance marked with tape on the floor
chair rise test | pre 16-week intervention
  The chair rise test is completed on a standard chair and provides information related to lower limb strength and agility. Subjects will be asked to stand up and sit down 5 times as fast as they can. Differences can be used descriptively but no definitive conclusions related to changes in fitness level can or will be made.
chair rise test | post 16-week intervention
  The chair rise test is completed on a standard chair and provides information related to lower limb strength and agility. Subjects will be asked to stand up and sit down 5 times as fast as they can. Differences can be used descriptively but no definitive conclusions related to changes in fitness level can or will be made.
Hand use | pre 16-week intervention
  An administrator capture whether or not the subject used their hands. (yes/no).
Physical Fitness Assessment (height) | post 16-week intervention
  subject's height will be taken using a wall-mounted stadiometer and weight will be taken using a medical-grade scale.
Resting Metabolic Rate | pre 16-week intervention
  Resting Metabolic Rate (RMR) will be measured using the CardioCoach or ReeVue (KORR Medical Technologies, Salt Lake City, UT). An RMR measurement uses oxygen consumed at rest to determine a person's caloric requirements for weight loss or maintenance
4-meter timed walk test | post 16-week intervention
  The 4-meter timed walk test will be used to measure normal gait speed and provide an approximate measure of physical functioning and level of deconditioning. The subject will be instructed to walk at their normal pace through a hallway that has a 4-meter distance marked with tape on the floor
Hand use | post 16-week intervention
  An administrator capture whether or not the subject used their hands. (yes/no).
Hand Dynamometer assessment | pre 16-week intervention
  provides a measure of upper body strength. The subject will be asked to squeeze as hard as he/she can and then relax. The average score of the three trials will be compared to the data norms. A dynamometer provides objective grip strength data. Males normally can generate about 46 kg of force, and females about 23 kg.
Hand Dynamometer assessment | post 16-week intervention
  provides a measure of upper body strength. The subject will be asked to squeeze as hard as he/she can and then relax. The average score of the three trials will be compared to the data norms. A dynamometer provides objective grip strength data. Males normally can generate about 46 kg of force, and females about 23 kg.
level of physical activity over the past 7 days | pre 16-week intervention
  Participants will also be asked 11 questions related to the frequency and amount of time spent in vigorous physical activity, moderate physical activity, walking, and sitting over the past 7 days.
level of physical activity over the past 7 days | post 16-week intervention
  Participants will also be asked 11 questions related to the frequency and amount of time spent in vigorous physical activity, moderate physical activity, walking, and sitting over the past 7 days.
Barratt's Impulsivity Scale (BIS-11), Inhibitory Control subscale | pre 16-week intervention
  a self-report questionnaire assessing the personality trait of impulsiveness. The scale includes 30 items covering attention, motor, and non-planning impulsiveness; only the Inhibitory Control subscale will be used for the purpose of this study - on a scale of "1" to "4": 1) rarely/never, 2) occasionally, 3) often, and 4) almost always/always
Urgency, Premeditation, Perseverance, and Sensation Seeking (UPPS) Impulsive Behavior Scale | pre 16-week intervention
  a self-report questionnaire assessing the personality trait of impulsiveness. The 45-item scale measures premediation, urgency, sensation-seeking, and perseverance; only the urgency subscale will be used for the purpose of the study - The Scale is not considered a measure of trait impulsivity, rather, the scales reflect distinct personality traits that lead to impulsive-type behavior. Participants are asked to consider acts/incidents during the last 6 months when rating their behavior and attitudes on a 4-point scale, in which 1-Agree strongly, 2-Agree some, 3-Disagree some, 4-Disagree strongly.The UPPS-P Negative Urgency scale (this is the only subscale on the UPPS we will be using) is a 12-item Likert-type scale to measure one's tendency to act rashly in response to intense negative mood states. It is a continuous scale, with higher scores meaning more negative urgency.
Posttraumatic Stress Disorder Checklist (PCL-5) | pre 16-week intervention
  is a 20 item self-report measure that assesses the DSM-5 symptoms of PTSD and is a commonly used tool to screen subjects for PTSD. Subjects rate each item from 1 ("not at all") to 5 ("extremely") to indicate the degree to which they have been bothered by that particular symptom over the past month.0 = Not at all 1 = A little bit 2 = Moderately 3 = Quite a bit 4 = Extremely Tally up score, total possible score range is 0-80. Score of >31 is considered significant for possible PTSD, <31 is considered non-significant for possible PTSD
Weight Control History | pre 16-week intervention
  Participants will also be asked questions related to their history of attempting to control their weight, including their weight at age 18, weight approximately 1 year ago, whether or not they have attempted to lose weight in the past year, and information related to their past 3 attempts at weight loss. Gathering this data for descriptive purposes, there is no "outcome," form of scoring, or analysis that will take place with this information.
Modified Yale Food Addiction Scale 2.0 (mYFAS 2.0) | week 1 post start of study
  an abbreviated, 13-item version of the Yale Food Addiction Scale 2.0 (YFAS 2.0). The mYFAS 2.0 has one question to assess each of the 11 DSM-5 diagnostic criteria for substance-use disorders, plus 2 questions to assess clinically significant distress and impairment. The modified versions of the YFAS perform similarly on psychometric indicators as the full versions of the scale and are useful brief assessment tool for food addiction.
Modified Yale Food Addiction Scale 2.0 (mYFAS 2.0) | week 5 post start of study
  an abbreviated, 13-item version of the Yale Food Addiction Scale 2.0 (YFAS 2.0). The mYFAS 2.0 has one question to assess each of the 11 DSM-5 diagnostic criteria for substance-use disorders, plus 2 questions to assess clinically significant distress and impairment. The modified versions of the YFAS perform similarly on psychometric indicators as the full versions of the scale and are useful brief assessment tool for food addiction.
Modified Yale Food Addiction Scale 2.0 (mYFAS 2.0) | week 9 post start of study
  an abbreviated, 13-item version of the Yale Food Addiction Scale 2.0 (YFAS 2.0). The mYFAS 2.0 has one question to assess each of the 11 DSM-5 diagnostic criteria for substance-use disorders, plus 2 questions to assess clinically significant distress and impairment. The modified versions of the YFAS perform similarly on psychometric indicators as the full versions of the scale and are useful brief assessment tool for food addiction.
Modified Yale Food Addiction Scale 2.0 (mYFAS 2.0) | week 15 post start of study
  an abbreviated, 13-item version of the Yale Food Addiction Scale 2.0 (YFAS 2.0). The mYFAS 2.0 has one question to assess each of the 11 DSM-5 diagnostic criteria for substance-use disorders, plus 2 questions to assess clinically significant distress and impairment. The modified versions of the YFAS perform similarly on psychometric indicators as the full versions of the scale and are useful brief assessment tool for food addiction.

SECONDARY OUTCOMES:
Dutch Eating Behavior Questionnaire (DEBQ) Excluding the restraint subscale | pre 16 week intervention
  The 33 question's scale ranges from 1 (never) to 5 (very often).with higher scores indicating greater endorsement of the eating behavior
Dutch Eating Behavior Questionnaire (DEBQ) Excluding the restraint subscale | post 16 week intervention
  The 33 question's scale ranges from 1 (never) to 5 (very often).with higher scores indicating greater endorsement of the eating behavior
Eating Disorder Examination - Questionnaire Short (EDE-QS) | pre 16 week intervention
  self-report measure assessing maladaptive eating behaviors. The questionnaire consists of 12 questions about eating behaviors in order to assess disordered eating behaviors - Scores on each item range from "0" to "6", with higher scores indicating higher symptom levels with higher scores indicating greater endorsement of the eating behavior
Eating Disorder Examination - Questionnaire Short (EDE-QS) | post 16 week intervention
  self-report measure assessing maladaptive eating behaviors. The questionnaire consists of 12 questions about eating behaviors in order to assess disordered eating behaviors - Scores on each item range from "0" to "6", with higher scores indicating higher symptom levels with higher scores indicating greater endorsement of the eating behavior
Eating Disorder Diagnostic Scale (EDDS) Restraint Subscale | pre 16 week intervention
  self-report measure assessing maladaptive eating behaviors consisting of 22 questions related to anorexia nervosa, bulimia nervosa, and binge-eating disorder - seven-point scale, ranging from 0 (not at all) to 6 (extremely)
Eating Disorder Diagnostic Scale (EDDS) Restraint Subscale | post 16 week intervention
  self-report measure assessing maladaptive eating behaviors consisting of 22 questions related to anorexia nervosa, bulimia nervosa, and binge-eating disorder - seven-point scale, ranging from 0 (not at all) to 6 (extremely)

CONTACTS AND LOCATIONS:
Overall Officials: Shenelle Edwards-Hampton, PhD, Principal Investigator — Wake Forest Health Sciences
Locations (1):
- Wake Forest Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes

DOCUMENTS (1):
  • Informed Consent Form (2023-03-22): https://cdn.clinicaltrials.gov/large-docs/43/NCT04373343/ICF_000.pdf